CLINICAL TRIAL: NCT04066179
Title: Efficacy of Monotherapy vs Combination Therapy of Corticosteroids With GCSF in Severe Alcoholic Hepatitis Patients -A Randomized Controlled Trial.
Brief Title: Efficacy of Monotherapy vs Combination Therapy of Corticosteroids With GCSF in Severe Alcoholic Hepatitis Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-AH-03
Record Dates: First submitted 2019-08-14; First posted 2019-08-26 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-08

CONDITIONS: Alcoholic Hepatitis
MeSH Terms: conditions — Hepatitis, Alcoholic | interventions — Granulocyte Colony-Stimulating Factor; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Prednisolone+G-CSF (Experimental): Prednisolone 40 mg/day for initial 7 days G-CSF300 microgram daily for 7 days
  Interventions: Drug: Gcsf; Drug: Prednisolone
- Prednisolone (Active Comparator): Prednisolone 40 mg/day for 7 days
  Interventions: Drug: Prednisolone
- Granulocytes-Colony Stimulating Factor (Experimental): Granulocytes-Colony Stimulating Factor 300 mcg for 7 days followed by 300 mcg every 3 days
  Interventions: Drug: Gcsf

INTERVENTIONS:
Drug: Gcsf — Granulocytes-Colony Stimulating Factor 300 mcg for 7 days followed by 300 mcg every 3 days
  Arms: Granulocytes-Colony Stimulating Factor; Prednisolone+G-CSF
Drug: Prednisolone — Prednisolone 40 mg for initial 7 days
  Arms: Prednisolone; Prednisolone+G-CSF

SUMMARY:
The patients of Severe Alcoholic Hepatitis (SAH) will be included in study based on inclusion and exclusion criteria. The patients will be then randomized in 3 groups for therapy. They will receive either steroid or Granulocyte-Colony Stimulating Factor (GCSF) or both. They will be followed for atleast 90 days for improvements in symptoms and various predefined parameters. Primary outcome will be improvement in survival at 90 Days. Patients will be monitored at every follow up for disease progression and complications of therapy. The study results will be analyzed for differences in survival rate and complications in different groups to propose new therapeutic guideline in SAH patients.

ELIGIBILITY:
Inclusion Criteria:

* Severe alcoholic hepatitis patients [Maddrey's score > 32] aged between 18 to 65 years.

Exclusion Criteria:

* Presence of active infections
* Acute Gastrointestinal bleed
* Hepatorenal syndrome
* Patient unwilling
* Discriminant Function >90
* Autoimmune hepatitis
* Hepatitis B, Hepatitis C, Human immunodeficiency Virus cases
* Pregnancy
* Hemophagocytic lymphohistiocytosis (HLH)
* Hb<8 and baseline White Blood Cell>25000

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2019-09-07 (Estimated); Primary Completion 2021-02-27 (Estimated); Study Completion 2021-02-27 (Estimated)

PRIMARY OUTCOMES:
increase in Survival at 90 days in all the groups. | 90 days

SECONDARY OUTCOMES:
Improvement in CTP (Child-Pugh Score) in all the groups. | Day 28
  CTP- Child-Turcotte-Pugh score ranges from 5 to 15, lowest is best and highest is worst.
Improvement in CTP (Child-Pugh Score) in all the groups. | Day 180
  CTP- Child-Turcotte-Pugh score ranges from 5 to 15, lowest is best and highest is worst.
Improvement in MELD (Model for End Stage Liver Disease) in all the groups. | Day 28
  A disease severity scoring system for adults with liver disease, designed to improve the organ allocation in transplantation based on the severity of liver disease rather than the length of time on the waiting list. A MELD score is a number that ranges from 6 to 40, based on lab tests.
Improvement in MELD (Model for End Stage Liver Disease) in all the groups. | Day 180
  A disease severity scoring system for adults with liver disease, designed to improve the organ allocation in transplantation based on the severity of liver disease rather than the length of time on the waiting list. A MELD score is a number that ranges from 6 to 40, based on lab tests.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No